CLINICAL TRIAL: NCT00921804
Title: A Phase IIa, Double-blind, Double-Dummy, Placebo-controlled, Active-controlled, Randomized, Parallel-Group Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of AZD8529 in Adult Schizophrenia Patients
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of AZD8529 in Adult Schizophrenia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1960C00004
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Hallucinations; Paranoia; Inpatient schizophrenia clinical trial
MeSH Terms: conditions — Schizophrenia; Hallucinations; Paranoid Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): AZD8529 40 mg
  Interventions: Drug: AZD 8529; Drug: Placebo to match risperidone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo to match AZD8529; Drug: Placebo to match risperidone
- 3 (Other): Risperidone 4 mg (2mg on Day 1)
  Interventions: Drug: Risperidone; Drug: Placebo to match AZD8529

INTERVENTIONS:
Drug: AZD 8529 — 40mg oral daily capsule administered as a single dose in the morning for 28 days
  Arms: 1
Drug: Risperidone — 4mg (2mg on Day 1) oral daily capsule administered as a single dose in the evening for 28 days
  Other Names: Risperdal
  Arms: 3
Drug: Placebo to match AZD8529 — Placebo to match AZD8529 administered as a daily capsule in the morning for 28 days during the treatment period and also during the 3-7 day washout or run-in period
  Arms: 2; 3
Drug: Placebo to match risperidone — Placebo to match risperidone administered as a daily capsule in the evening for 28 days during the treatment period and also during the 3-7 day washout or run-in period
  Arms: 1; 2

SUMMARY:
The purpose of this study is to determine whether treatment with daily oral dose of AZD8529 40 mg administered over 28 days is safe, well tolerated and improves main symptoms of schizophrenia in adult schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient will need to read, understand and sign an informed consent prior to any study specific procedures
* Patient will have certain schizophrenia symptoms deemed by the investigator as appropriate for the study entry

Exclusion Criteria:

* Patients will be excluded based on recent history of significant illness or current disease as assessed by the investigator during screening process (based on physical examination, laboratory studies and electrocardiogram studies)
* Patients will be excluded if urine drug screen test show positive results
* Smoking of more than 2 packs of cigarettes a day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
PANSS Total Score | Prior to randomization (screening, admission to washout/run in, baseline) and Days 8, 15, 22, and 28

SECONDARY OUTCOMES:
PANSS Positive, Negative, and General Psychopathology Subscale Scores | Prior to randomization (screening, admission to washout/run in, baseline) and Days 8, 15, 22, and 28
CGI-S | Prior to randomization (screening, admission to washout/run in, baseline) and Days 8, 15, 22, and 28
Vital signs measurements, body weight, physical exam, clinical laboratory evaluations, ECGs, Extrapyramidal Symptoms, suicidal symptoms, cognition and incidence of adverse events | Prior to randomization (screening, admission to washout/run in, baseline) and Days 1, 8, 15, 22, and 28

CONTACTS AND LOCATIONS:
Overall Officials: Robert, Litman, M.D, Principal Investigator — CBH Health9605 Medical Center Drive Suite 270Rockville, MD, 20850; Mark Smith, Study Director — AstraZeneca1800 Concord PikeWilmington, DE, 19850
Locations (3):
- United States (3):
  - Research Site, Garden Grove, California
  - Research Site, Glendale, California
  - Research Site, Rockville, Maryland